CLINICAL TRIAL: NCT00604214
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Study of Drotrecogin Alfa (Activated) Administered as a Continuous 96-hr Infusion to Adult Patients With Septic Shock
Brief Title: Efficacy and Safety of Drotrecogin Alfa (Activated) in Adult Patients With Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11940; F1K-MC-EVDP (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-24; First posted 2008-01-30 (Estimated); Results first posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-08

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — drotrecogin alfa activated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drotrecogin alfa (activated) (Experimental)
  Interventions: Drug: Drotrecogin alfa (activated)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drotrecogin alfa (activated) — 24 microgram/kilogram/hour, intravenous, 96 hours (hr)
  Other Names: LY203638; Xigris
  Arms: Drotrecogin alfa (activated)
Drug: Placebo — 0.9% sodium chloride, intravenous, 96 hours
  Arms: Placebo

SUMMARY:
The purpose of this placebo-controlled study is to determine if drotrecogin alfa (activated) treatment provides significant mortality reduction improvement in patients with septic shock compared with placebo treatment in patients receiving the current standard of care for septic shock. This study will also assess the effectiveness of drotrecogin alfa (activated) in reducing 28-day mortality in patients with septic shock and concomitant severe protein C deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must have evidence of infection
* Must have systemic inflammatory response syndrome (SIRS)
* Must have vasopressor-dependent septic shock

Exclusion Criteria:

* Have received vasopressor therapy (at any dose) for greater than 24 hours prior to the start of study drug
* Have sepsis-induced organ dysfunction for greater than 36 hours prior to the start of the study drug infusion
* Have single organ dysfunction and recent surgery (within 30 days of study entry)
* Have had surgery performed within the 12-hour period immediately preceding the study drug infusion, or are postoperative with evidence of active bleeding, or have planned or anticipated surgery during the infusion period
* Are not expected to survive 28 days given their preexisting uncorrectable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1696 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (149):
- United States (23):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hazard, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
- Australia (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Epping, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria
- Belgium (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., LiÃ¨ge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottignies
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roeselare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilrijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yvoir
- Brazil (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joinville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Londrina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sao Jose Rio Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., SÃ£o Paulo
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thunder Bay, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrook, Quebec
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hradec Králové
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pilsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ústí nad Labem
- Finland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jyväskylä
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lahti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seinäjoki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
- France (23):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Argenteuil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bobigny
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Kremlin-Bicêtre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poissy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pringy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Michel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aachen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
- Italy (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varese
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tlalpan
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ede
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
- New Zealand (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auckland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grafton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Spain (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcalá de Henares
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burgos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Palmas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murcia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tortosa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valladolid
- Switzerland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lugano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sankt Gallen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- United Kingdom (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelmsford, Essex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edinburgh, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chichester, West Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London

REFERENCES:
- [Derived] Povoa P, Salluh JI, Martinez ML, Guillamat-Prats R, Gallup D, Al-Khalidi HR, Thompson BT, Ranieri VM, Artigas A. Clinical impact of stress dose steroids in patients with septic shock: insights from the PROWESS-Shock trial. Crit Care. 2015 Apr 28;19(1):193. doi: 10.1186/s13054-015-0921-x. PMID 25928214
- [Derived] Ranieri VM, Thompson BT, Barie PS, Dhainaut JF, Douglas IS, Finfer S, Gardlund B, Marshall JC, Rhodes A, Artigas A, Payen D, Tenhunen J, Al-Khalidi HR, Thompson V, Janes J, Macias WL, Vangerow B, Williams MD; PROWESS-SHOCK Study Group. Drotrecogin alfa (activated) in adults with septic shock. N Engl J Med. 2012 May 31;366(22):2055-64. doi: 10.1056/NEJMoa1202290. Epub 2012 May 22. PMID 22616830
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Drotrecogin Alfa (Activated): 24 microgram/kilogram/hour, intravenous, 96 hours
Period: Baseline to Day 28
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Started | 851 | 845
Received Study Drug | 833 | 833
Completed | 623 | 632
Not Completed | 228 | 213
Not completed — Death | 223 | 202
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 3 | 7
Period: Day 29 to Day 90
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Started | 623 | 632
Completed | 555 | 553
Not Completed | 68 | 79
Not completed — Death | 64 | 67
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 0 | 6
Period: Day 91 to Day 180
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Started | 555 | 553
Completed | 529 | 521
Not Completed | 26 | 32
Not completed — Death | 19 | 23
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drotrecogin Alfa (Activated) | Placebo | Total
Number analyzed (Participants) | 851 | 845 | 1696
Age Continuous [Mean (Standard Deviation); unit: years] | 63.42 (15.42) | 62.70 (16.41) | 63.06 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 379 | 739
  Male | 491 | 466 | 957
Race/Ethnicity, Customized [Number; unit: participants]
  Aboriginal/Torres Strait Islander | 2 | 6 | 8
  African | 30 | 27 | 57
  Caucasian | 740 | 721 | 1461
  East Asian/Pacific | 21 | 10 | 31
  Hispanic | 21 | 32 | 53
  Native American | 3 | 4 | 7
  West Asian (Indian Subcontinent) | 34 | 45 | 79
Region of Enrollment [Number; unit: participants]
  Portugal | 3 | 5 | 8
  United States | 78 | 82 | 160
  Finland | 45 | 42 | 87
  Spain | 87 | 84 | 171
  Switzerland | 8 | 10 | 18
  United Kingdom | 44 | 49 | 93
  Italy | 54 | 53 | 107
  India | 40 | 41 | 81
  France | 235 | 229 | 464
  Czech Republic | 30 | 24 | 54
  Mexico | 7 | 7 | 14
  Canada | 36 | 43 | 79
  Brazil | 18 | 18 | 36
  Belgium | 69 | 70 | 139
  Australia | 36 | 28 | 64
  Netherlands | 15 | 15 | 30
  Germany | 22 | 23 | 45
  New Zealand | 24 | 22 | 46
Primary Site of Infection [Number; unit: participants]
  Abdomen | 263 | 246 | 509
  Blood | 40 | 25 | 65
  Bone | 2 | 2 | 4
  Central Nervous System | 11 | 9 | 20
  Head | 2 | 3 | 5
  Heart | 3 | 3 | 6
  Lung | 369 | 375 | 744
  Other | 11 | 17 | 28
  Pleura | 2 | 5 | 7
  Reproductive Tract | 2 | 2 | 4
  Skin or Skin Structure | 48 | 45 | 93
  Urinary Tract | 97 | 112 | 209
  Unknown | 1 | 1 | 2
Cardiovascular Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing cardiovascular dysfunction. There were 12 participants in drotrecogin alfa (activated) and 14 participants in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 3.91 (0.32) | 3.89 (0.35) | 3.90 (0.33)
Respiratory Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing respiratory dysfunction. There were 35 participants in drotrecogin alfa (activated) and 34 participants in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 2.78 (1.07) | 2.74 (1.08) | 2.76 (1.08)
Renal Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing renal dysfunction. There were 12 participants in drotrecogin alfa (activated) and 17 participants in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 1.67 (1.33) | 1.60 (1.34) | 1.63 (1.33)
Coagulation Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating worsening coagulopathy (decreasing platelet counts). There were 11 participants in drotrecogin alfa (activated) and 17 participants in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 0.76 (0.97) | 0.71 (0.96) | 0.74 (0.96)
Liver Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing liver dysfunction. There were 61 participants in drotrecogin alfa (activated) and 70 participants in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 0.55 (0.85) | 0.53 (0.88) | 0.54 (0.87)
Acute Physiology and Chronic Health Evaluation II (APACHE II) Score [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II (APACHE II) score is a severity-of-disease classification system. Scores range from 0 to 71. Higher scores correspond to more severe disease and a higher risk of death. There were 4 participants in drotrecogin alfa (activated) and 1 participant in placebo who were unspecified and were not included in the calculation of mean and standard deviation.
  units on a scale | 25.17 (8.06) | 25.45 (8.14) | 25.31 (8.10)

OUTCOME MEASURES:

1. Primary Outcome: 28-Day All-Cause Mortality
Description: Expressed as percentage of participants who died from any cause at Day 28 endpoint.
Time Frame: Day 28
Population: All randomized participants with known mortality status at Day 28.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 846 | 834
percentage of participants | 26.4 | 24.2
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; The study was planned to have 80% power to detect a 20% relative risk reduction in 28-day all-cause mortality in drotrecogin alpha (activated) compared to placebo. The final power was 75% because of the lower than anticipated placebo mortality; Test type: Superiority or Other; p = 0.313, Chi-squared — No adjustment for multiple comparisons; Risk Ratio (RR) = 1.088, 95% CI 2-sided [0.923 to 1.283]

2. Secondary Outcome: 28-Day All-Cause Mortality in Participants With Severe Protein C Deficiency
Description: Expressed as percentage of participants who died from any cause at Day 28 endpoint. Participants with severe protein C deficiency are those who had a protein C level ≤ half the lower limit of normal (LLN) (≤40%).
Time Frame: Day 28
Population: All randomized participants with severe protein C deficiency at Baseline with known mortality status at Day 28.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 342 | 331
percentage of participants | 28.7 | 30.8
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.540, Chi-squared — No adjustments for multiple comparisons; Risk Ratio (RR) = 0.930, 95% CI 2-sided [0.737 to 1.173]

3. Secondary Outcome: Average Cardiovascular Sequential Organ Failure Assessment (SOFA) Score Day 1 Through Day 28
Description: Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing cardiovascular dysfunction. A non-surviving participant receives a score of 4 (worst score) for the day of death and every day thereafter.
Time Frame: Day 1 through Day 28
Population: All randomized participants with any post-baseline data on Day 1 through Day 28. For those days when a participant is alive, but no data are available, last observation carried forward (LOFC) is used to impute the missing data. A non-surviving participant receives a score of 4 (worst score) for the day of death and every day thereafter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 837 | 828
units on a scale | 1.92 (1.31) | 1.84 (1.31)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.181, ANOVA — No adjustments for multiple comparisons

4. Secondary Outcome: Average Respiratory Sequential Organ Failure Assessment (SOFA) Score Day 1 Through Day 28
Description: Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing respiratory dysfunction. A non-surviving participant receives a score of 4 (worst score) for the day of death and every day thereafter.
Time Frame: Day 1 through Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 817 | 806
units on a scale | 2.31 (1.05) | 2.29 (1.05)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.733, ANOVA — No adjustments for multiple comparisons

5. Secondary Outcome: Average Renal Sequential Organ Failure Assessment (SOFA) Score Day 1 Through Day 28
Description: Scores range from 0 (normal) to 4 (organ failure) with an increasing score indicating increasing renal dysfunction. A non-surviving participant receives a score of 4 (worst score) for the day of death and every day thereafter.
Time Frame: Day 1 through Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 836 | 827
units on a scale | 1.38 (1.42) | 1.28 (1.40)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.122, ANOVA — No adjustments for multiple comparisons

6. Secondary Outcome: 90-Day Mortality
Description: Expressed as percentage of participants who died from any cause at Day 90 endpoint.
Time Frame: Day 90
Population: All randomized participants with known mortality status at Day 90.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 842 | 822
percentage of participants | 34.1 | 32.7
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.556, Chi-squared — No adjustments for multiple comparisons; Risk Ratio (RR) = 1.042, 95% CI 2-sided [0.909 to 1.193]

7. Secondary Outcome: 180-Day Mortality
Description: Expressed as percentage of participants who died from any cause at Day 180 endpoint.
Time Frame: Day 180
Population: All randomized participants with known mortality status at Day 180.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 835 | 813
percentage of participants | 36.6 | 35.9
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.758, Chi-squared — No adjustments for multiple comparisons; Risk Ratio (RR) = 1.020, 95% CI 2-sided [0.898 to 1.160]

8. Secondary Outcome: Median Survival Time
Time Frame: Day 180
Population: All randomized participants excluding those with unknown mortality status at Day 180.
Measure: Median (Full Range); unit: days
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 835 | 813
days | NA [NA to NA] — Median value was not calculated due to less than 50% of participants reaching mortality endpoint at Day 180. | NA [NA to NA] — Median value was not calculated due to less than 50% of participants reaching mortality endpoint at Day 180.

9. Secondary Outcome: EuroQoL Questionnaire-5 Dimensions (EQ-5D) Visual Analog Scale (VAS) Scores at Baseline, Days 28, 90 and 180
Description: EQ-5D VAS assesses caregiver's impression of participant's overall health state. Scores range from 0 (worst health state) to 100 (best health state), with higher scores indicating a better health state.
Time Frame: Baseline and Days 28 and 90 and 180
Population: All randomized participants with EQ-5D VAS data at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 851 | 845
units on a scale
  Baseline (n=685, 679) | 54.21 (26.99) | 54.37 (27.95)
  Day 28 (n=500, 476) | 54.78 (23.46) | 55.24 (22.89)
  Day 90 (n=474, 469) | 64.41 (21.00) | 65.18 (20.15)
  Day 180 (n=456, 443) | 68.94 (20.19) | 69.08 (20.50)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.788, ANOVA — P-value is for Baseline, unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.730, ANOVA — P-value is for Day 28, unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.662, ANOVA — P-value is for Day 90, unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.846, ANOVA — P-value is for Day 180, unadjusted for multiple comparisons

10. Secondary Outcome: EuroQoL Questionnaire-5 Dimensions (EQ-5D) Total Scores at Baseline, Days 28, 90 and 180
Description: The EQ-5D is used to assess participant's overall health. Consists of 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has 3 severity levels (no, some, severe problems). Calculated from EQ-5D, total scores (United States [US] Index Score) range from 0 (worst quality of life) to 1.00 (best quality of life).
Time Frame: Baseline and Days 28 and 90 and 180
Population: All randomized participants with EQ-5D total score data at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 851 | 845
units on a scale
  Baseline (n=702, 705) | 0.60 (0.35) | 0.60 (0.35)
  Day 28 (n=509, 486) | 0.51 (0.33) | 0.53 (0.33)
  Day 90 (n=480, 473) | 0.71 (0.27) | 0.71 (0.28)
  Day 180 (n=458, 448) | 0.77 (0.23) | 0.76 (0.25)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.697, ANOVA — P-value is for Baseline, unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.306, ANOVA — P-value is for Day 28, unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.645, ANOVA — P-value is for Day 90, unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.690, ANOVA — P-value is for Day 180, unadjusted for multiple comparisons

11. Secondary Outcome: Quality of Life Short Form-12 (SF-12) Scores at Baseline, Days 28, 90 and 180
Description: SF-12 was used as an instrument to measure participants' physical wellbeing (physical component) and mental wellbeing (mental component). Scores for each component range from 0-100, with 0= lowest wellbeing, and 100=highest wellbeing.
Time Frame: Baseline and Days 28 and 90 and 180
Population: All randomized participants with SF-12 score data at the specified time points.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 851 | 845
units on a scale
  Physical Component at Baseline (n=683, 696) | 39.14 (12.04) | 39.22 (12.10)
  Physical Component at Day 28 (n=484, 465) | 31.14 (10.29) | 31.13 (9.84)
  Physical Component at Day 90 (n=474, 459) | 38.09 (11.17) | 40.03 (11.23)
  Physical Component at Day 180 (n=450, 444) | 42.26 (10.80) | 41.59 (11.28)
  Mental Component at Baseline (n=683, 696) | 45.44 (13.07) | 46.03 (12.88)
  Mental Component at Day 28 (n=484, 465) | 40.57 (13.12) | 41.45 (12.59)
  Mental Component at Day 90 (n=474, 459) | 47.53 (12.08) | 48.52 (12.36)
  Mental Component at Day 180 (n=450, 444) | 50.42 (11.50) | 50.55 (11.70)
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.482, ANOVA — P-value is for physical component at Baseline, unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.584, ANOVA — P-value is for physical component at Day 28, unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.164, ANOVA — P-value is for physical component at Day 90, unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.666, ANOVA — P-value is for physical component at Day 180, unadjusted for multiple comparisons
Statistical Analysis 5: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.786, ANOVA — P-value is for mental component at Baseline, unadjusted for multiple comparisons
Statistical Analysis 6: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.160, ANOVA — P-value is for mental component at Day 28, unadjusted for multiple comparisons
Statistical Analysis 7: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.696, ANOVA — P-value is for mental component at Day 90, unadjusted for multiple comparisons
Statistical Analysis 8: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Analysis on ranked data; Test type: Superiority or Other; p = 0.966, ANOVA — P-value is for mental component at Day 180, unadjusted for multiple comparisons

12. Other Pre Specified Outcome: Percentage of Participants With Serious Bleeding Events Within System Organ Class Any Time From Baseline Through Day 28
Description: Percentage of participants who experienced serious bleeding events are reported by System Organ Class (SOC) term based on MedDRA 14.0. For a bleeding to qualify as a serious event, it would have to meet the standard definition of a serious adverse event or be a central nervous system bleeding or a bleeding event that lead to administration of ≥3 units packed red blood cells/day for 2 consecutive days.
Time Frame: Baseline through Day 28
Population: Participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 833 | 833
percentage of participants
  with ≥1 event | 2.4 | 2.8
  Gastrointestinal Disorders | 1.1 | 0.7
  Injury, Poisoning And Procedural Complications | 0 | 0.6
  Nervous System Disorders | 0.4 | 0.4
  Renal And Urinary Disorders | 0.1 | 0
  Respiratory, Thoracic And Mediastinal Disorders | 0.4 | 0.4
  Vascular Disorders | 0.5 | 1.0
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.758, Fisher Exact — P-value is for participants with ≥1 event. No adjustments for multiple comparisons

13. Secondary Outcome: Percentage of Participants Discontinued Due to Adverse Events Any Time From Baseline Through Day 28 Endpoint
Time Frame: Baseline through Day 28
Population: Participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Number analyzed (Participants) | 833 | 833
percentage of participants | 4.4 | 3.0
Statistical Analysis 1: Comparison: Drotrecogin Alfa (Activated) vs Placebo; Test type: Superiority or Other; p = 0.154, Fisher Exact — Unadjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28
Arm/Group | Drotrecogin Alfa (Activated) | Placebo
Serious Adverse Events (participants affected / at risk) | 119/833 | 96/833
Other Adverse Events (participants affected / at risk) | 151/833 | 119/833
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drotrecogin Alfa (Activated) (N=833) | Placebo (N=833)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 2 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (6) | 1 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 13 (15) | 8 (8)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 4 (5) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (4) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Pupils unequal (Eye disorders) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 3 (5)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 3 (4) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (3) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (2) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (3) | 2 (2)
Rectal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2)
Device dislocation (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Idiosyncratic drug reaction (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (3) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (7) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (2) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 0 (0)
Colon gangrene (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (2)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 1 (2) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (10) | 3 (3)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia staphylococcal (Infections and infestations) | 2 (3) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Superinfection bacterial (Infections and infestations) | 1 (3) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Urosepsis (Infections and infestations) | 4 (6) | 2 (5)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (5) | 2 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Oxygen saturation decreased (Investigations) | 1 (2) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 2 (3)
Cerebral haemorrhage (Nervous system disorders) | 2 (4) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (4) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (3) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (5) | 4 (5)
Neuroleptic malignant syndrome (Nervous system disorders) | 0 (0) | 1 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (3)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal infarct (Renal and urinary disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (2) | 1 (3)
Haemorrhage (Vascular disorders) | 1 (3) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 2 (2)
Intra-abdominal haemorrhage (Vascular disorders) | 2 (2) | 3 (5)
Peripheral ischaemia (Vascular disorders) | 2 (4) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 3 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drotrecogin Alfa (Activated) (N=833) | Placebo (N=833)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 1 (3)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (21) | 9 (17)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 3 (9)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (4)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 8 (16) | 5 (9)
Atrial thrombosis (Cardiac disorders) | 1 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (7)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Deafness bilateral (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 4 (10) | 3 (4)
Scleral haemorrhage (Eye disorders) | 1 (3) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 6 (9) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 6 (7)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 3 (5) | 6 (7)
Mouth haemorrhage (Gastrointestinal disorders) | 3 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bloody discharge (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 9 (9) | 4 (6)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Mucosal haemorrhage (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (4)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 (9) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 11 (18) | 2 (5)
Alanine aminotransferase increased (Investigations) | 1 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0)
Occult blood positive (Investigations) | 2 (3) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 1 (1)
Prothrombin time prolonged (Investigations) | 2 (5) | 0 (0)
Prothrombin time shortened (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 11 (12) | 9 (18)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal infarct (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Scrotal haematocoele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Arterial thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (2) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 10 (26) | 5 (17)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2) | 2 (2)
Intra-abdominal haematoma (Vascular disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 2 (4)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (3)
Phlebitis (Vascular disorders) | 0 (0) | 1 (3)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (4)
Thrombophlebitis (Vascular disorders) | 1 (1) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 4 (10)
Thrombosis (Vascular disorders) | 1 (4) | 3 (6)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 1 (4)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the site PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo. An independent Steering Committee responsible for data analyses and publications did not have an embargo.